CLINICAL TRIAL: NCT01400607
Title: Randomized Controlled Trial to Evaluate the Efficacy of a Neocartilage Implant in the Management of ICRS Grade 3 to 4 Articular Cartilage Lesions of the Knee
Brief Title: Neocartilage Implant to Treat Cartilage Lesions of the Knee
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: ISTO Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISTO NEO-01-09-01
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2016-09

CONDITIONS: Articular Cartilage Disorder; Degeneration; Articular Cartilage; Chronic Cartilage Injury; Acute Cartilage Injury; Defect of Articular Cartilage
Keywords: cartilage; knee surgery; cartilage injury; knee pain; cartilage repair; cartilage damage; cartilage lesion; cartilage defect; articular cartilage lesion; articular cartilage defect; juvenile; cells; ISTO Technologies; Neocartilage; RevaFlex
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neocartilage Implant (Active Comparator): Neocartilage Implant surgically implanted and affixed to subchondral bone using commercial fibrin during mini-open knee arthrotomy.
  Interventions: Biological: Neocartilage Implant/DeNovo® ET (Engineered Tissue Graft)
- Microfracture (Other): Standard of care cartilage repair technique.
  Interventions: Other: Microfracture

INTERVENTIONS:
Biological: Neocartilage Implant/DeNovo® ET (Engineered Tissue Graft) — The Neocartilage Implant is a cartilage repair technology cultured from juvenile human cartilage cells.
  Other Names: RevaFlex
  Arms: Neocartilage Implant
Other: Microfracture — Marrow stimulation using the microfracture technique; performed arthroscopically
  Other Names: marrow stimulation
  Arms: Microfracture

SUMMARY:
ISTO Technologies, Inc. is proposing a clinical study with 225 subjects, to establish the safety and efficacy of the Neocartilage Implant for the treatment of ICRS Grade 3 and 4 articular cartilage lesions of the knee compared to microfracture treatment.

DETAILED DESCRIPTION:
In the United States alone, more than 500,000 cartilage lesions per year require some treatment to reduce pain, restore joint mobility, and prevent further damage caused by the progression of osteoarthritis. The lack of effective cartilage repair approaches or products for restoration of defective articular cartilage to its native, hyaline morphology only continues to exacerbate the incidence of osteoarthritis as these initial defects enlarge and degrade over a 10 to 20 year period. The repair of cartilage, especially in the knee, remains a formidable clinical challenge. Regenerative medicine approaches to cartilage repair have only begun to be explored as possible options and there is a clear trend toward biological solutions for the repair and regeneration of damaged or diseased articular cartilage. The study was designed to compare how well the Neocartilage Implant works against the microfracture therapy, a widely used and accepted cartilage repair therapy. Data to be collected include Pain and Function in Daily Living scores, symptoms, Function in Sports and Recreation, and Knee Related Quality of Life. Additionally, MRI and X-rays will be collected to evaluate the cartilage repair progress. These assessments will be used through the five years of post-operative follow-up.

ELIGIBILITY:
Inclusion Criteria:

Generally, the following inclusion criteria must be met, however, this is not a complete list.

* Male or Female between the ages of 18 and 60
* (1) or (2) articular cartilage lesions of the distal femur ranging in no more than 5 cm2 each
* Ipsilateral knee compartment has intact menisci (or meniscectomized remnant with > 5mm wide rim) and stable ligaments in the affected knee
* 3 months out from initiation of conservative non-surgical management (e.g.hyaluronic acid injection, activity modification) or previous minimal surgical intervention (e.g., arthroscopic lavage, debridement) or 12 months out from marrow stimulation for this condition

Exclusion Criteria:

Generally, if a potential participant meets any of the following criterions, they will not be eligible for this study. Additionally, more criteria will be evaluated to confirm eligibility as this list is not a complete list of criteria.

* Osteoarthritis
* Rheumatoid arthritis
* History of septic or reactive arthritis
* Gout or a history of gout or pseudo-gout in the affected knee
* Osteochondritis dissecans or osteochondral lesions of the knee with bone loss > 6mm deep
* Bipolar articular cartilage involvement (or kissing lesions) of the ipsilateral compartment (i.e., > than ICRS Grade 2 on the opposing articular surface)
* Associated damage to the underlying subchondral bone requiring an osteochondral graft
* Is pregnant or breast-feeding
* Has a BMI > 35 (kg/m2)
* Has prior total meniscectomy of either knee
* Has received, within the past three months, intra-articular hyaluronic acid therapy, or steroid therapy
* Has more than two clinically relevant chondral lesion(s) on the index knee

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Scores (KOOS) | 36 months
  Knee Injury and Osteoarthritis Outcomes Scores (KOOS) Pain and Function in Daily Living (ADL) subscales.

SECONDARY OUTCOMES:
IKDC Knee Examination | Baseline, 6 week, 6, 12, 18, 24 months and annually through 5 years
Subject reported questionnaires | Baseline, 6 week, 6, 12, 18, 24 months and annually through 5 years
  Various questionnaires are required to be completed by the subject before and after treatment throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Purcell, Study Director — ISTO Technologies, Inc.
Locations (9):
- United States (9):
  - Kerlan Jobe Orthopaedic Clinic, Los Angeles, California
  - Santa Monica Orthopaedic & Sports Medicine Group, Santa Monica, California
  - Rush University Medical Center, Chicago, Illinois
  - Hospital for Special Surgery -Sports Medicine and Shoulder Service, New York, New York
  - Insall Scott Kelly Institute for Orthopaedics & Sports Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Sports Medicine Center, Columbus, Ohio
  - The Hawkins Foundation, Greenville, South Carolina
  - The Methodist Hospital Research Institute, Houston, Texas